CLINICAL TRIAL: NCT00138086
Title: Targeted Intensification by a New Preparative Regimen for Patients With Low-Grade B-Cell Lymphoma Utilizing Standard-Dose Yttrium-90 Ibritumomab Tiuxetan (Zevalin) Radioimmunotherapy (RIT) Combined With High-Dose Beam Followed by Autologous Stem Cell Transplantation (ASCT)
Brief Title: Yttrium-90 Ibritumomab Tiuxetan (Zevalin) With BEAM in Relapsed Low Grade B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z-BEAM
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: B-Cell Lymphoma
Keywords: lymphoma; chemotherapy; Zevalin ( Yttrium-90 Ibritumomab Tiuxetan)
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma | interventions — ibritumomab tiuxetan

INTERVENTIONS:
Drug: Zevalin plus BEAM

SUMMARY:
The objective of this study is to evaluate the efficacy and the safety of Zevalin-BEAM preparative regimen before autologous stem cell transplantation (ASCT) as measured by the event free survival (EFS).

The goal is to obtain a 15% increase of EFS at 2 years.

DETAILED DESCRIPTION:
The indolent course of the low-grade B-cell lymphoma is thus characterized by multiple remissions and relapses with ever-shortening "time to progression" intervals, and by ultimately becoming refractory to treatment. In this situation of recurrences, intensive therapy including high-dose chemotherapy or chemo-radiotherapy followed by autologous hematopoietic stem cell transplantation appears as a therapeutic option. With the use of peripheral blood stem cell, the autologous stem cell transplantation (ASCT) procedure has become easier and cheaper, and it has a mortality rate of below 5% and manageable morbidity. EBMT registry data or institution driven studies have shown an improvement in event free survival when compared to chemotherapy in relapsing patients. Recently Schouten et al reported in a randomized study a significant benefit in survival for patients submitted in relapse to ASCT. Consolidation with ASCT has been studied in first line treatment and showed a significant improvement in survival in one randomized study. BEAM regimen is a referent high-dose chemotherapy used in intensive therapy followed by ASCT in the treatment of malignant lymphoma. It could therefore be considered for patients with indolent lymphoma if it could be shown to improve survival. In most studies the conditioning regimen was associating chemotherapy and Total Body Irradiation (TBI) for indolent lymphoma as it is very sensitive to even low dose of radiotherapy. TBI however is time consuming and technically not available in all transplant centers and associated with some long term toxicities; a search for more specific targeted irradiation has been a goal for several years.

Recently, a new preparative regimen for older patients with aggressive CD20-positive B-cell lymphoma utilizing standard-dose 0.4 mCi/kg 90Y ibritumomab tiuxetan combined with high-dose BEAM followed by ASCT showed a CR rate of 92% with a follow-up of 9 months. Finally, high-dose radioimmunotherapy with 90Y ibritumomab tiuxetan and high-dose cyclophosphamide/etoposide followed by ASCT for poor-risk or relapsed B-cell NHL have been reported, with a 2-year DFS of 80%. The use of conventional dose of Yttrium did not need heavy radioprotection procedures, and can be widely distributed in transplant centers.

Overall toxicities were comparable to standard autologous transplantation conditioning regimens, and the combined treatment was well tolerated. The hematological reconstitution after transplantation occurred without delay, except in two cases than in control-based high-dose chemotherapy alone population. Mucositis and neutropenic fever were reported without increase of severity. Nonhematological adverse events have been observed, three interstitial pneumonitis, mild abnormalities on liver or kidney function tests, except one case of veno-occlusive disease, and 4 fatal infection (disseminated aspergillosis with a brain abscess, streptococcal sepsis, staphylococcal sepsis, and disseminated varicella zoster).

Therefore, all these data support a phase II trial evaluating efficacy and toxicities in patients with low grade B-Cell lymphoma of a new preparative regimen combining a standard dose 90Y ibritumomab tiuxetan and high-dose BEAM chemotherapy followed by ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Patients with pathologically proven at relapse, low grade B-cell lymphoma CD20- positive (World Health Organization [WHO] classification):

  * Marginal zone;
  * Lymphocytic; or
  * Follicular.
* In relapse after complete remission (CR), less than partial remission (PR) or partial response (maximum of 3 lines of treatment)
* Previously treated with chemotherapy regimen with or without rituximab
* With a chemo-sensitive disease using salvage therapy
* Eligible for autologous stem cell transplantation
* ECOG performance status 0 to 2
* Minimum life expectancy of 3 months
* Negative HIV, hepatitis B virus (HBV) and hepatitis C virus (HCV) serologies < 4 weeks (except after vaccination)
* Signed informed consent form

Exclusion Criteria:

* Histological transformation in diffuse large cell from a low grade B-cell lymphoma
* Prior transplantation
* Contraindication to any drug contained in the chemotherapy regimens
* Large bone marrow irradiation > 40%
* Bone marrow infiltration > 25%
* Lack of sufficient autologous stem cells for transplantation
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study
* Any serious active disease or co-morbid medical condition (according to the investigator's decision and information provided in the Investigational Drug Brochure [IDB])
* Poor bone marrow reserve as defined by neutrophils < 1.5 G/l or platelets < 100 G/l, unless related to bone marrow infiltration
* Poor renal function (creatinine level > 2.5 maximum normal level) unless abnormalities are related to the lymphoma
* Poor hepatic function (total bilirubin level > 30 mmol/l, transaminases > 2.5 maximum normal level) unless abnormalities are related to the lymphoma
* Any history of cancer during the last 5 years, with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma
* Presence of anti-murine antibody (HAMA) reactivity
* Known hypersensitivity to murine antibodies or proteins
* Pregnant women
* Adult patients unable to give informed consent because of intellectual impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2005-03; Study Completion 2009-03

PRIMARY OUTCOMES:
EFS (event free survival)

SECONDARY OUTCOMES:
Overall response rate (ORR)
Toxicities, transplant related mortality at 1 and 2 years
Hematological reconstitution after ASCT and 1 year
Time to progression or relapse, disease free survival for complete responders after ASCT, overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gisselbrecht, MD PHD, Principal Investigator — Lymphoma Study Association
Locations (9):
- Groupe d'Etude des Lymphomes de l'adulte, Mont-Godinne, Belgium
- France (7):
  - Hôpital Henri Mondor, Créteil
  - Hématologie CHU de Lille, Lille
  - Institut Curie, Paris
  - Hôpital Saint Louis, Paris
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - Institut Gustave Roussy, Villejuif
- Schweirische Arbeitsgruppe fur klinische Krebsforschung, Lausanne, Switzerland

REFERENCES:
- [Background] Brice P, Simon D, Bouabdallah R, Belanger C, Haioun C, Thieblemont C, Tilly H, Harousseau JL, Doyen C, Martin C, Brousse N, Solal-Celigny PH; Groupe d'Etude des Lymphomes de l'Adulte (GELA). High-dose therapy with autologous stem-cell transplantation (ASCT) after first progression prolonged survival of follicular lymphoma patients included in the prospective GELF 86 protocol. Ann Oncol. 2000 Dec;11(12):1585-90. doi: 10.1023/a:1008399623564. PMID 11205467
- [Background] Mills W, Chopra R, McMillan A, Pearce R, Linch DC, Goldstone AH. BEAM chemotherapy and autologous bone marrow transplantation for patients with relapsed or refractory non-Hodgkin's lymphoma. J Clin Oncol. 1995 Mar;13(3):588-95. doi: 10.1200/JCO.1995.13.3.588. PMID 7884420
- [Background] Witzig TE, White CA, Gordon LI, Wiseman GA, Emmanouilides C, Murray JL, Lister J, Multani PS. Safety of yttrium-90 ibritumomab tiuxetan radioimmunotherapy for relapsed low-grade, follicular, or transformed non-hodgkin's lymphoma. J Clin Oncol. 2003 Apr 1;21(7):1263-70. doi: 10.1200/JCO.2003.08.043. PMID 12663713
- [Background] Fung HC, Forman SJ, Nademanee A, Molina A, Yamauchi D, Speilberger R, Kogut N, Sahebi F, Parker P, Rodriguez R, Krishnan A, Popplewell L, Wong J, and Raubitschek A. A new preparative regimen for older patients with aggressive CD20-positive B-cell lymphoma utilizing standard-dose Yttrium-90 Ibritumomab Tiuxetan (Zevalin) radioimmunotherapy (RIT) combined with high-dose BEAM followed by autologous hematopoietic cell transplantation (AHCT) : targeted intensification without increased transplant-related toxicity. Blood 2003, forty-fifth annual meeting of the American Society of Hematology, abstract 870.
- [Background] Nademanee A, Forman SJ, Molina A, Kogut N, Fung HC, Yamauchi D, Anderson A-L, Smith D, Liu AN, and Raubitschek A. High-dose radioimmunotherapy with yttrium 90 (90Y) ibritumomab tiuxetan with high-dose etoposide (VP-16) and cyclophosphamide (CY) followed by autologous hematopoietic cell transplantation (AHCT) for poor-risk or relapsed B-cell non-Hodgkin's lymphoma (NHL): update of a phase I/II trial. J Clin Oncol 2004, fortieth annual meeting of the American Society of Clinical Oncology, abstract 6504.
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In french) — http://www.gela.org